CLINICAL TRIAL: NCT03056430
Title: Neuroanatomical and Functional Changes in Response to an Intensive Balance Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Center for Neurodegenerative Diseases (DZNE) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: MD038
Record Dates: First submitted 2016-12-27; First posted 2017-02-17 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2018-03

CONDITIONS: Spatial Orientation; Balance
Keywords: MRI, Neuroplasticity, Balance, Spatial orientation, Hippocampus, Slacklining
MeSH Terms: conditions — Orientation, Spatial

STUDY DESIGN:
Intervention Model Description: Repeated-measures, 2 groups * 2 timepoints
Oversight: Data Monitoring Committee: No

ARMS (2):
- Training Group 1 (Experimental): Slackline training
  Interventions: Behavioral: Training
- Training Group 2 (Experimental): Slackline training
  Interventions: Behavioral: Training

INTERVENTIONS:
Behavioral: Training

SUMMARY:
The purpose of this study is to determine whether intensive slackline training improves spatial orientation abilities, balancing skills and causes neuroplasticity in related brain cortical regions.

ELIGIBILITY:
Inclusion Criteria:

* No previous slacklining or related experience, 18-30 years of age, good or corrected to good vision

Exclusion Criteria:

* Musculoskeletal and nervous system injuries/diseases that significantly reduce one's ability to perform slacklining training, systemic diseases (cardiovascular, gastrointestinal, metabolic...)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline at 1 and 3 months in Balance Tests score | Baseline, 1 month post-test, 3 months post-test
Change from Baseline at 1 and 3 months in Spatial Orientation Tests score | Baseline, 1 month post-test, 3 months post-test
Change from Baseline at 1 and 3 months in voxel-wise morphometric brain analysis | Baseline, 1 month post-test, 3 months post-test

CONTACTS AND LOCATIONS:
Overall Officials: Notger Müller, Prof. Dr., Principal Investigator — German Center for Neurodegenerative Diseases (DZNE)
Locations (1):
- DZNE, Magdeburg, Saxony-Anhalt, Germany

IPD SHARING:
Plan to Share IPD: No